CLINICAL TRIAL: NCT03253900
Title: Changes of Biomechanical Parameters During Race Simulation Rowing - The Effect of (In)Stability of the Simulator
Brief Title: Rowing Biomechanics - Effects of (In)Stability and Fatigue
Acronym: RowBio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Responsible Party: Principal Investigator, Nejc Sarabon, Assoc. Prof. Dr. Sc., University of Primorska
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UP-FVZ-RowingBiomechanics
Record Dates: First submitted 2017-08-05; First posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Healthy
Keywords: wobble board; slides; rowing stroke; rowing biomechanics; power output

STUDY DESIGN:
Intervention Model Description: All participants in the study will complete the measurements for all the three rowing interventions; in a random order.
Masking Description: The investigator who processed the acquired data was blinded for rowing interventions and subject information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): A group of rowers to be administered to intervention on a Stable rowing simulator, a Slides based rowing simulator or a Tilt board based rowing simulator.
  Interventions: Device: Stable rowing simulator; Device: Slides based rowing simulator; Device: Tilt board based rowing simulator

INTERVENTIONS:
Device: Stable rowing simulator — a standard stable/fixed rowing simulator
Device: Slides based rowing simulator — a slides based rowing simulator, i.e. horizontal plane unstable
Device: Tilt board based rowing simulator — a tilt board based rowing simulator; i.e. frontal plane unstable

SUMMARY:
Rowing simulators are frequently used by rowers, when on-water training is impossible or limited. While such devices are highly valuable to maintain rowers' fitness, a concern was raised about extensive simulator usage. It was postulated that it could lead to technique alterations due to different biomechanical properties compared to on-water rowing. Slide-based rowing simulators were designed to better simulate on-water conditions.

The main aim of the study was to compare the differences in various kinematic and kinetic parameters during a short (20 s) all-out rowing bout and during a 2000-m simulated race, to get a better insight into how different rowing simulator designs affect biomechanics of rowing.

Three different rowing simulators were used in this study: (1) a standard stable/fixed rowing simulator, (2) a slides based rowing simulator, i.e. horizontal plane unstable, and (3) a tilt board based rowing simulator; i.e. frontal plane unstable.

The investigators hypothesised that rowing on different simulators will elicit different biomechanics, including forces, power output, arm and seat movement velocity and amplitude.

Each of the participants completed the tests in all three interventions on separate sessions; random order of interventions. The three sessions took place 7-10 days apart. During each session, the participants completed the all-out 20-s trial first, then the simulated 2000-m race. The aforementioned biomechanical parameters were tracked throughout the trials to be compared between interventions later.

DETAILED DESCRIPTION:
The measurements will take place at University of Primorska (Koper, Slovenia) and the subjects will be recruited in close collaboration with Rowing Club Piran. Crossover study design will be used. Each participant will be asked to come for three visits that will be scheduled 7-10 days apart. Prior to measurements onset, the whole protocol will be explained to the participant.

Measurement procedure:

* 15-min warm-up
* 20-s maximal (all-out) rowing
* 5-minute break
* 2000-m simulated race

After both trials, blood lactate will be measured. Blood sample will be taken at the the earlobe by a qualified medical personnel.

Maximal performance test: The participant will perform a 20-s interval with maximal effort. The main aim of the measurement is to record the maximal exerted force and power. The custom adapted device (Concept 2 Rowing Simulator) records the positions (seat and handle) and force (legs push and handle pull), which enables for further calculations of segmental and common kinematics and dynamics parameters.

Race simulation: the participant will complete the 2000-m simulated race and will be instructed to aim for the best results. The same measurements as in the maximal performance test will be performed. Wireless heart rate monitor will be used to record the heart frequency throughout the trial.

Equipment:

The custom adapted rowing simulator (Concept 2) allows for the measurements of stoke forces and consequently power outputs, seat and handle velocity, and seat and handle amplitudes. Signals will be transferred to central unit, amplified and converted, and stored on a personal computer.

The interventions (i.e. the studied rowing conditions) will be as follows:

* a standard stable/fixed rowing simulator,
* a slides based rowing simulator, i.e. horizontal plane unstable, and
* a tilt board based rowing simulator; i.e. frontal plane unstable.

ELIGIBILITY:
Inclusion Criteria:

* Competitive rowers with at least 4 years of experience
* Completed the physical examination at sports physician
* Parental consent for underage participants

Exclusion Criteria:

* Injury in last 12 months
* Any health issues that may be exacerbated by interventions

Ages: 15 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Rowing performance | Three sessions, with randomized order of ergometers (7-10 days apart)
  Rowing biomechanics on different rowing simulators.

SECONDARY OUTCOMES:
Arm velocity | At the onset of test, at the finish and at the three points in between (at 500, 1000 and 1500 meters of the simulated race) - ref. POM: sessions 7-10 days apart.
  Change of the average velocity of arm movement through the rowing stroke.
Seat velocity | At the onset of test, at the finish and at the three points in between (at 500, 1000 and 1500 meters of the simulated race) - ref. POM: sessions 7-10 days apart.
  Change of the average velocity of the seat movement through the rowing stroke.
Arm force | At the onset of test, at the finish and at the three points in between (at 500, 1000 and 1500 meters of the simulated race) - ref. POM: sessions 7-10 days apart.
  Change of the average arm force through the rowing stroke.
Handle amplitude | At the onset of test, at the finish and at the three points in between (at 500, 1000 and 1500 meters of the simulated race) - ref. POM: sessions 7-10 days apart.
  Change of the average handle through the rowing stroke.
Leg force | At the onset of test, at the finish and at the three points in between (at 500, 1000 and 1500 meters of the simulated race) - ref. POM: sessions 7-10 days apart.
  Change of the average leg force through the rowing stroke.
Seat amplitude | At the onset of test, at the finish and at the three points in between (at 500, 1000 and 1500 meters of the simulated race) - ref. POM: sessions 7-10 days apart.
  Change of the average amplitude of the seat movement through the rowing stroke.
Lactate | Before and immediately after the test, ref. POM: sessions 7-10 days apart. .
  Change in blood lactate concentration

IPD SHARING:
Plan to Share IPD: Undecided